CLINICAL TRIAL: NCT03669666
Title: Role of Phase Contrast Magnetic Resonance in Regurgitant Valvular Heart Diseases
Brief Title: Phase Contrast in Valvular Heart Disease
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdulrahman Emam Eldeen, principal investigator, Assiut University
Other Study IDs: PC-CMR-VHDs
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Valvular Heart Disease (Aortic and Mitral Valves)
Keywords: valvular heart disease; ejection fraction
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: 10 normal healthy subjects are conducted for cardiac magnetic resonance imaging examination
- case group: 25 patients with valvular heart disease diagnosed clinically and by echocardiography are conducted for cardiac magnetic resonance imaging examination

SUMMARY:
The ability to quantify flow directly using through-plane phase contrast velocity mapping is a unique advantage of cardiovascular magnetic resonance and does not rely on the calculation from complex equations as echocardiography.

The aim s is to study the role of cardiac MRI in the evaluation of valvular heart disease through quantification of the impact of valvular lesions upon cardiac function by accurate estimation of the left ventricular ejection fraction

DETAILED DESCRIPTION:
Valvular heart disease is common and increases with age. In the past, valvular heart disease was typically caused by rheumatic heart disease, which remains a significant public health burden in developing countries. In industrialized nations, however, the rheumatic diseases has fallen substantially and valvular heart disease is now mainly degenerative in origin.

Valvular heart disease encompasses a number of common cardiovascular conditions that account for 10% to 20% of all cardiac surgical procedures.

Clinical examination is not a reliable guide to diagnosis or severity. This gap in the clinical valvular heart disease and the late presentation of many with severe disease emphasizes the importance of quantitative, high-quality cardiac imaging.

Imaging needs to assess: 1) valve morphology to determine the etiology and suitability for invasive intervention; 2) hemodynamic severity; 3) remodeling of the left ventricle and right ventricle; 4) involvement of the aorta and 5) the prediction of adverse cardiovascular events.

A number of imaging modalities are currently available to evaluate valvular heart disease in a comprehensive manner allowing correct assessment of both valve morphology and function. Doppler-echocardiography is the most frequently used tool for this purpose because it is cost-effective, widely available and, in the majority of the cases, provides sufficient information for clinical patient management and possible surgical planning.

For a long time, cardiac catheterization and invasive angiography have been regarded as the "gold standard". However, this invasive approach exposes patients to radiation and iodinated contrast media, carrying the non-negligible risk of life-threatening complications but nonetheless far from optimal especially regarding the precise quantification of valvular regurgitation.

Due to considerable improvements in hard- and software design in the last decade, magnetic resonance imaging has claimed its role as a central player in a large variety of cardiac diseases offering unique information about the mechanism of valve disease, quantifying the severity of disease, and discerning the consequences of the lesions including the effects on left ventricular volume, left ventricular systolic function, and left atrial volumes. Because of both its high accuracy and reproducibility, magnetic resonance imaging has become the preferred imaging modality in an increasing number of clinical trials. Also in the field of valvular heart disease, considerable progress has been achieved.

Today, cardiovascular magnetic resonance has a number of unique advantages over other imaging modalities. It provides a view of the entire heart without limitations from inadequate imaging windows or body habitus. Additionally, in some patients, information from clinical history and physical examination or other diagnostic tests may be discordant with echocardiographic findings where there is a significant clinical role for cardiovascular magnetic resonance. cardiovascular magnetic resonance also can obtain imaging data in any imaging plane prescribed by the scan operator, which makes it ideal for accurate investigation of all cardiac valves: aortic, mitral, pulmonic, and tricuspid. It can be considered an excellent adjunct to echocardiography for investigating patients with valve disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically diagnosed valvular heart disease and confirmed by echocardiography

Exclusion Criteria:

* Patients with known contraindication to MRI including the presence of paramagnetic
* Surgical clips, or pacemakers
* Severely ill patients
* Claustrophobic or restless subjects
* Patients with arrhythmia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted on 35 subjects including 25 patients with reversed cardiac hemodynamics and 10 age- and sex-matched healthy adult controls with no clinically or echocardiographically detected cardiac abnormalities. The 25 patients have been diagnosed clinically and by echocardiography to have valvular heart disease of different aetiologies (14 rheumatics, 5 ischemic, 6 non-ischemic cardiomyopathies).
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
measurement of ejection fraction | 1 day
  measurement of ejection fraction via estimation of stroke volume divided by end diastolic volume of the left ventricle

CONTACTS AND LOCATIONS:
Locations (1):
- abdulrahman Emam, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iung B, Baron G, Butchart EG, Delahaye F, Gohlke-Barwolf C, Levang OW, Tornos P, Vanoverschelde JL, Vermeer F, Boersma E, Ravaud P, Vahanian A. A prospective survey of patients with valvular heart disease in Europe: The Euro Heart Survey on Valvular Heart Disease. Eur Heart J. 2003 Jul;24(13):1231-43. doi: 10.1016/s0195-668x(03)00201-x. PMID 12831818
- [Background] Maganti K, Rigolin VH, Sarano ME, Bonow RO. Valvular heart disease: diagnosis and management. Mayo Clin Proc. 2010 May;85(5):483-500. doi: 10.4065/mcp.2009.0706. PMID 20435842
- [Background] Chambers JB, Myerson SG, Rajani R, Morgan-Hughes GJ, Dweck MR. Multimodality imaging in heart valve disease. Open Heart. 2016 Mar 8;3(1):e000330. doi: 10.1136/openhrt-2015-000330. eCollection 2016. PMID 26977308
- [Background] Simpson IA, Sahn DJ. Quantification of valvular regurgitation by Doppler echocardiography. Circulation. 1991 Sep;84(3 Suppl):I188-92. PMID 1884485
- [Background] Myerson SG. Heart valve disease: investigation by cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2012 Jan 19;14(1):7. doi: 10.1186/1532-429X-14-7. PMID 22260363